CLINICAL TRIAL: NCT00557882
Title: A Randomized Clinical Trial of Vaginal Mesh for Anterior Prolapse
Brief Title: Efficacy Study of Vaginal Mesh for Anterior Prolapse
Acronym: VAMP-A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-336
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Vaginal Prolapse; Uterine Prolapse; Cystocele; Pelvic Organ Prolapse
Keywords: prolapse; uterus; mesh; bladder
MeSH Terms: conditions — Uterine Prolapse; Cystocele; Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mesh (Active Comparator): Vaginal reconstructive surgery with synthetic polypropylene mesh
  Interventions: Device: synthetic polypropylene mesh
- no mesh (Active Comparator): Vaginal reconstructive surgery without mesh
  Interventions: Device: synthetic polypropylene mesh

INTERVENTIONS:
Device: synthetic polypropylene mesh — Mesh used will be synthetic monofilament polypropylene. In this trial, patients in the experimental group will undergo interpositional multi-armed mesh placement using trocars for transobturator +/- ischioanal fossa placement at the level of the ischial spine.

SUMMARY:
The primary aim of this double-blind, randomized clinical trial (RCT) is to test the hypothesis that the addition of a standardized technique of interpositional synthetic polypropylene mesh placement improves the one-year outcome of vaginal reconstructive surgery for anterior prolapse compared to traditional vaginal reconstructive surgery without mesh.

DETAILED DESCRIPTION:
Multiple vaginal, abdominal and laparoscopic procedures have been described for surgical correction of pelvic support problems. However, conventional pelvic reconstructive surgeries have been associated with a 20-30% prolapse recurrence rate. The anterior vaginal wall is the site most often recognized as the area of vaginal prolapse recurrence. Minimally invasive surgical procedures using mesh have rapidly developed in the field of pelvic floor reconstruction in an attempt to improve surgical cure rates. Unfortunately, safety and efficacy data have lagged behind the technical advancements.

This trial will randomize women with advanced anterior wall prolapse to two treatment arms: vaginal reconstructive surgery with mesh and vaginal reconstructive surgery without mesh. The primary outcome is cure of anterior wall prolapse at one year. Secondary outcomes are cure of apical and posterior wall prolapse, quality-of-life measures and complication rates. Patients will be approached for recruitment only after they have made the decision to undergo vaginal surgery for anterior prolapse. The patient and examiner will be blinded to the surgical treatment assignment. Interim measurement of primary and secondary outcomes will be conducted three months post-operatively. Additional follow-up will be conducted at one-year intervals subsequent to the expected one-year endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. women age > 21
2. diagnosed with stage II-IV vaginal prolapse who desire reconstructive surgery
3. available for 12 months of follow-up
4. able to complete study questionnaires and assessments.
5. available for 12 months follow-up

Exclusion Criteria:

1. Uterus in place.
2. No anterior vaginal prolapse.
3. Medical contraindications, e.g. current urinary tract, vaginal or pelvic infection, history of pelvic irradiation, history of lower urinary tract malignancy, chronic steroid use or a compromised immune system.
4. Current intermittent self catheterization.
5. Pregnancy or desire for future fertility.
6. Presence of an adnexal or ovarian mass.
7. Shortened vagina.
8. Other laparoscopic or abdominal/pelvic surgery in the past 3 months.*
9. Known neurologic or medical condition affecting bladder function, e.g. multiple sclerosis, spinal cord injury.
10. Need for surgery requiring an abdominal incision.
11. <12 months post-partum. (Enrollment can be deferred until time requirement has been met).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew I Sokol, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Wahington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- See also: Click clinical trials for more information about this study " A Randomized Clinical trial of Vaginal Mesh for Prolapse" — http://medstarresearch.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mesh | no Mesh
Started | 32 | 33
Completed | 27 | 33
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesh | no Mesh | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.8) | 63.5 (8.9) | 63.94 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure for Objective Treatment Success is Anterior Prolapse, Point Ba at Stage 0 or 1 (Defined as Maximal Descent of the Anterior Wall to Greater Than 1 cm Above the Hymen) at One Year.
Time Frame: 1 year
Population: NIH optimal prolapse cure (Pelvic Organ Prolapse Quantifications System (POP-Q) stage <1)
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh | no Mesh
Number analyzed (Participants) | 32 | 33
Participants | 12 | 10

ADVERSE EVENTS:
Arm/Group | Mesh | no Mesh
All-Cause Mortality (participants affected / at risk) | 1/32 | 1/33
Serious Adverse Events (participants affected / at risk) | 5/32 | 0/33
Other Adverse Events (participants affected / at risk) | 4/32 | 1/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesh (N=32) | no Mesh (N=33)
mesh erosion (Injury, poisoning and procedural complications) | 5 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesh (N=32) | no Mesh (N=33)
cystotomy (Renal and urinary disorders) | 2 | 0
Febrile Illness (General disorders) | 1 | 1
Postoperative blood transfusion (General disorders) | 1 | 0 — Postoperative blood transfusion for participant with concurrent hystorectomy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No